CLINICAL TRIAL: NCT00735813
Title: A Randomised Study of Taurolock for the Locking of Tunneled Central Venous Catheters in Children With Malignant Diseases.
Brief Title: Taurolidine Lock Solution in the Prevention of Catheter Related Bacteremia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: Danish Child Cancer Foundation (Other); TauroPharm (Industry)
Responsible Party: Principal Investigator, Mette Møller Handrup, MD, PhD, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17344
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Bacteremia; Neoplasms
Keywords: Catheterization, Central; Catheterization, Peripheral; Infection; Methods; Sepsis; Microscopy, Electron, Scanning; Sonication; Taurolidine; Catheters, Indwelling; Pediatrics
MeSH Terms: conditions — Bacteremia; Neoplasms; Infections; Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Tunneled central venous catheters locked with Taurolock
  Interventions: Device: Taurolock
- B (Active Comparator): Tunneled central venous catheter locked with heparin
  Interventions: Device: Heparin

INTERVENTIONS:
Device: Taurolock — When not in use the childrens tunneled central venous catheters are locked with the liquid Taurolock instead of heparin.
  Arms: A
Device: Heparin — When not in use the childrens tunneled central venous catheters are locked with heparin
  Arms: B

SUMMARY:
Children with cancer need a long term tunnelled central venous catheter (TCVC) for the entire duration of their treatment. TCVCs are locked with heparin when not in use. The most frequent complications of long term TCVC are catheter related blood steam infections. Taurolock is a new lock that is claimed to prevent the formation of luminal biofilm in TCVCs and has been demonstrated to eradicate infected CVCs. In this study the investigators will compare TCVCs locked with heparin with TCVCs locked with Taurolock. Hypothesis: Taurolock will diminish the number of CRBSI in children with cancer compared with children with heparin lock of their CVC.

DETAILED DESCRIPTION:
The most frequent complications of long term TCVC are catheter related blood steam infections(CRBSI)often caused by microorganisms located in the biofilm formed on the inner surface of the TCVC after a short time. CRBSI may be lifethreatening, will need long term intravenous broad spectrum antibiotic therapy possibly combined with intraluminal antibiotic lock therapy. In spite of this CRBSI may often lead to the premature removal of the TCVC.

Several methods to prevent the occurrence of intraluminal microbial colonization have been investigated with no single method standing out as the optimal one.

There is a need for a simple and safe method of reducing the occurrence of CRBSI in immunocompromised children receiving chemotherapy for malignant diseases. Various catheter lock solutions in stead of using heparin have been investigated in experimental models. Taurolidine is a chemically modified amino acid with broad spectrum antimicrobial activity in vitro. It is claimed to prevent the formation of luminal biofilm in TCVCs in a CVC model and it has been demonstrated to eradicate infected CVC in a three reports with a total of 18 patients.

In a 24 months study of routine use of Taurolidine 1,25%/Sodium-Citrate 4% (TaurolockTM) a reduction of gram-positive CVC associated infections was demonstrated. The findings were not statistically significant due to relatively few patients.

There is a need of a larger study with more patients receiving Taurolock for locking the TCVC between use in order to test for a significant reduction of the occurrence of CRBSI. Furthermore there is a need for an in vivo demonstration of the reduction of biofilm formation in TCVCs locked with taurolock compared with TCVCs locked with heparin.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0-17 years with malignant disease requiring a tunneled central venous catheter.

Exclusion Criteria:

* No written consent from child or parents

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 129 (Actual)
Dates: Start 2008-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Number of catheter related blood stream infections(CRBSI)in the Taurolock group vs the heparin group. Number of CRBSI/1000 CVC days in the Taurolock group vs the heparin group. Number of CVCs removed in the Taurolock group vs the heparin group | November 2010

SECONDARY OUTCOMES:
Biofilm formation in the CVCs treated with Taurolock compared with the biofilm formation in the CVCs treated with heparin | February 2010

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Schrøder, MD, Dr.med., Study Director — Aarhus Universityhospital, Skejby
Locations (1):
- Childrens Department of Oncology A4, Aarhus Universityhospital, Skejby, Århus N, Denmark

REFERENCES:
- [Background] Bradshaw JH, Puntis JW. Taurolidine and catheter-related bloodstream infection: a systematic review of the literature. J Pediatr Gastroenterol Nutr. 2008 Aug;47(2):179-86. doi: 10.1097/MPG.0b013e318162c428. PMID 18664870
- [Background] Betjes MG, van Agteren M. Prevention of dialysis catheter-related sepsis with a citrate-taurolidine-containing lock solution. Nephrol Dial Transplant. 2004 Jun;19(6):1546-51. doi: 10.1093/ndt/gfh014. Epub 2004 Feb 19. PMID 14993498
- [Background] Raad I, Hanna H, Maki D. Intravascular catheter-related infections: advances in diagnosis, prevention, and management. Lancet Infect Dis. 2007 Oct;7(10):645-57. doi: 10.1016/S1473-3099(07)70235-9. PMID 17897607
- [Background] O'Grady NP, Alexander M, Dellinger EP, Gerberding JL, Heard SO, Maki DG, Masur H, McCormick RD, Mermel LA, Pearson ML, Raad II, Randolph A, Weinstein RA; Healthcare Infection Control Practices Advisory Committee. Guidelines for the prevention of intravascular catheter-related infections. Infect Control Hosp Epidemiol. 2002 Dec;23(12):759-69. doi: 10.1086/502007. PMID 12517020
- [Background] Raad I, Hanna HA, Alakech B, Chatzinikolaou I, Johnson MM, Tarrand J. Differential time to positivity: a useful method for diagnosing catheter-related bloodstream infections. Ann Intern Med. 2004 Jan 6;140(1):18-25. doi: 10.7326/0003-4819-140-1-200401060-00007. PMID 14706968
- [Derived] Handrup MM, Moller JK, Schroder H. Central venous catheters and catheter locks in children with cancer: a prospective randomized trial of taurolidine versus heparin. Pediatr Blood Cancer. 2013 Aug;60(8):1292-8. doi: 10.1002/pbc.24482. Epub 2013 Feb 15. PMID 23417891
- See also: Related Info — http://www.taurolock.de